CLINICAL TRIAL: NCT00799786
Title: Building Better Caregivers Online
Brief Title: Building Better Caregivers Online: An Online Workshop for Caregivers of Those With Traumatic Brain Injury, Post Traumatic Stress Disorder, or Alzheimer's or Other Dementia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Kate R Lorig, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SU-11212008-1350; 40137
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Last update posted 2010-08-13 (Estimated); Status verified 2010-08

CONDITIONS: Dementia; Brain Injuries; Stress Disorders, Traumatic
MeSH Terms: conditions — Dementia; Brain Injuries; Stress Disorders, Traumatic

INTERVENTIONS:
Behavioral: Building Better Caregivers Online Workshop

SUMMARY:
The workshop is a 6-week online workshop for caregivers of people with traumatic brain injury, post traumatic stress disorder, or dementia. It is being conducted jointly by the Stanford Patient Education Research Center and the VA Greater Los Angeles Healthcare System and is supported by a grant from the Department of Veterans Affairs, Patient Care Services, Office of Care Management and Social Work.

The goal of the study is to determine whether an online caregiver education and support workshop can have lasting beneficial effects in helping caregivers improve their self-management of health skills, stress, and improve their caregiving abilities.

DETAILED DESCRIPTION:
The workshop is a 6-week online workshop for caregivers of people with traumatic brain injury, post traumatic stress disorder, or dementia. It is being conducted jointly by the Stanford Patient Education Research Center and the VA Greater Los Angeles Healthcare System and is supported by a grant from the Department of Veterans Affairs, Patient Care Services, Office of Care Management and Social Work.

The goal of the study is to determine whether an online caregiver education and support workshop can have lasting beneficial effects in helping caregivers improve their self-management of health skills, stress, and improve their caregiving abilities.

This study is designed to enroll 120 participants living in California, Hawaii or Southern Nevada. Your participation in the workshop is expected to last six weeks, and the study will last 1 year.

This workshop is aimed at helping you to better manage your own health and the demands placed on you because of caregiving.

With the moderators and other workshop participants, you will discuss:

* Stress reduction
* Goal setting
* Maintaining your health
* Dealing with difficult emotions
* Handling difficult behaviors
* Better decision making
* Communicating better with health care professionals
* Communicating better with your friends, family and coworkers

If you participate in the workshop, you will take it online with 20-25 other people like you who are caregivers for veterans with TBI, PTSD, or dementia, or are veterans giving care to someone with these disorders. Each week you will log on to the study web site at least three times for a total time per week of about 2 hours. The first time you log on each week should be on the first or second day of the workshop, but you may log on at any time you find convenient. You may log on as often as you wish and at any time during the week. There is no time when all of you must log on at the same time.

Each week, you will be asked to read material on line, to complete activities on the web site, to make and share an action plan (for something you choose each week), to share your caregiving-related problems with others in your group, and most important of all, to help and support other group members with your experiences and wisdom. You will participate by using an anonymous screen name, and none of the other workshop members will know your real name.

Everyone in the study will be asked to fill out 4 brief online questionnaires about your health, medical care, activities and mood. You will fill out one questionnaire now, one two months after the beginning of the workshop, and another one in six months, and one in one year. Each questionnaire will take about 30 minutes to complete. Shortly after the workshop, we may ask you to participate in an email discussion group designed to get your feedback about the workshop. For the follow up questionnaires at 2, 6 and 12 months after you start the workshop you will receive a $10 Amazon.com certificate for each questionnaire to compensate you for your time and effort.

ELIGIBILITY:
Inclusion Criteria:Any adult (18 and over) who provides caregiving services for at least 10 hours per week (counting direct caregiving and related activities) for a veteran with traumatic brain injury, post traumatic stress disorder, or dementia, or is a veteran giving care to someone with one of these disorders, and has access to the internet and an email account. A caregiver is defined as any relative, partner, friend or neighbor who has a significant personal relationship with and provides a broad range of assistance for an older person or an adult with a chronic or disabling condition. These individuals may be the sole caregiver or one of several that live with or separately from the person receiving care.

* Live in California
* Have access to the internet and an email account
* Able to read English Exclusion Criteria:Live outside of California, Hawaii or Southern Nevada, under 18 years of age, not have access to a computer and own emai

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
quality o flife, health status, and medical care utilization | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kate R Lorig, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Greater Los Angeles VA, Los Angeles, California
  - Stanford University School of Medicine, Stanford, California